CLINICAL TRIAL: NCT05414045
Title: Autologous Testicular Tissue Transplantation for Fertility Restoration
Brief Title: Autologous Testicular Tissue Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-477
Record Dates: First submitted 2022-02-17; First posted 2022-06-10 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Sickle Cell Thalassemia; Hematologic Diseases
MeSH Terms: conditions — Neoplasms; Hematologic Diseases

STUDY DESIGN:
Intervention Model Description: All eligible patients for the study will have the same treatment: autologous testicular tissue transplantation with testicular tissue containing spermatogonial stem cells frozen at pre-pubertal age. Transplantation will be performed subcutaneously in the scrotum and intra-testicular.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental)
  Interventions: Procedure: Autologous testicular tissue transplantation of prepubertal frozen testicular tissue

INTERVENTIONS:
Procedure: Autologous testicular tissue transplantation of prepubertal frozen testicular tissue — Freezing testicular tissue of prepubertal boys is a method for preserving spermatogonial stem cells (SSCs).
  If the patient has a childwish on adult age and in case no spermatozoa are found in the ejaculate, the investigators will perform autologous testicular tissue transplantation with the primary objective being to restore spermatogenesis and fertility.

SUMMARY:
Freezing testicular tissue of prepubertal boys is a method for preserving spermatogonial stem cells (SSCs) in case of imminent gonadotoxic treatment during childhood. In case of total azoospermia in adulthood and presence of a childwish, the investigators intend to perform the first in men autologous testicular tissue transplantation to restore fertility.

DETAILED DESCRIPTION:
Freezing testicular tissue of prepubertal boys is a method for preserving spermatogonial stem cells (SSCs). In 2002, the University hospital in Brussels (UZB) was the first hospital worldwide to offer testicular tissue cryobanking for fertility preservation in boys and ado-lescents. Since then, several other centers in Europe and USA have implemented similar fertility preservation programs. However, up till now, autologous transplantations of cryopreserved testicular tissue have not been performed yet.

As soon as a patient returns to the Centre for Reproductive Medicine at UZB with the request to transplant the preserved testicular tissue, the investigators will first analyse semen and blood. If spermatozoa are found in their semen, men can immediately enroll in standard care for natural conception, intra-uterine insemination (IUI), in-vitro fertilization (IVF) or intra-cytoplasmic injection (ICSI). However, in case no spermatozoa are found in the ejaculate the investigators intend to propose and eventually perform autologous testicular tissue transplantation with the primary objective being to restore spermatogenesis and fertility.

ELIGIBILITY:
The eligible patients opted as a prepubertal boy to enroll in the fertility preservation program and on the moment of cancer diagnosis or hematological disorder, their parents have agreed to cryopreserve testicular tissue for later autologous transplantation.

Inclusion Criteria:

* At least 18 years old
* Desire to become a parent at the moment of intake
* Stable relationship with a female partner and minimal one year cohabiting
* Age of female partner < 43 year
* Azoospermia on 2 semen analyses
* Normal standardised preliminary and preoperative bloodsampling results
* Complete remission of the oncological or hematological disease
* Approval of the treating oncologist or other specialist in case of non-oncological disease as reason for the testicular tissue preservation as a child
* Risk for presence of malignant cells in testicular tissue is negligible (according to multidisciplinary assessment)
* Presence of SSCs (positive MAGE staining) in one or two of the thawed fragments (If absence of SSCs in two of the thawed fragments, the case will be discussed multidisciplinary)
* Written informed consent for the transplantation of cryopreserved testicular tissue and follow-up after the procedure and of children born eventually after this procedure

Exclusion criteria:

* Risk for presence of malignant cells in the testicular tissue
* Contra-indication for surgery
* Contra-indication for pregnancy in the female partner
* BMI > 32
* Heavy smoking (≥10 cigarettes/day)
* Instable psychological condition

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male infertile survivors of childhood cancer or a hematological disease who underwent prepubertal testicular tissue cryopreservation in case of gonadotoxic treatment.
Enrollment: 5 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2030-07-29 (Estimated); Study Completion 2030-10-29 (Estimated)

PRIMARY OUTCOMES:
Restoration of spermatogenesis and fertility by performing an autologous testicular tissue transplantation. Primary endpoint is the presence of spermatozoa in the graft. | Graft-removal of intratesticular and intrascrotal grafts is planned 12 months after grafting.
  Freezing testicular tissue of prepubertal boys is a method for preserving spermatogonial stem cells (SSCs).
  If the patient has a childwish at adult age and in case no spermatozoa are found in the ejaculate, the investigators will perform autologous testicular tissue transplantation with the primary objective being to restore spermatogenesis and fertility.
  Grafting will be performed intra-testicular and intrascrotal for each patient. Grafts will be removed 12 months after grafting.
  Primary endpoint is the presence of spermatozoa in the grafted tissue. In the IVF laboratory mechanical mincing and enzymatic digestion will be performed on the tissue to find spermatozoa. If spermatozoa are present concentration and motility will be available.

SECONDARY OUTCOMES:
Histological study to define the optimal transplantation site | Graft-removal of intratesticular grafts and intrascrotal grafts are planned 12 months after initial grafting. Histological study will be performed 12 months after initial grafting
  The presence of sperm-generating stem cells, as well as their possible maturation to sperm cells will be evaluated through available and validated microscopic staining techniques applied to the testicular tissue. The maturity of other, non-sperm-generating testicular cells (Sertoli cells and Leydig cells) will also be evaluated. The results from tissue fragments transplanted to the testicle will be compared to the results from the tissue fragments transplanted to the scrotum. During the removal procedure of the transplanted fragments, a control biopsy (TESE) will be performed on the contra-lateral testicle (the one on which no transplantation was performed).
Imaging study | Each patient in the study will be followed-up after screening during a period of 12 months post-grafting on 3, 6, 9 and 12 months after initial grafting.
  The investigators will study the possibility of analyzing the growth of the transplanted fragments and the development of sperm cell production in these fragments by using ultrasound and Doppler techniques in a non-invasive way. Ultrasound will be performed 3, 6, 9 and 12 months after grafting. These findings will be compared to the findings of the semen and blood analysis and the clinical examination.
Endocrinological (hormonal) study | Each patient in the study will be followed-up after screening during a period of 12 months post-grafting on 3, 6, 9 and 12 months after initial grafting.
  The investigators plan a follow-up of the functionality of the transplanted tissue by performing blood analyses with LH (IU/L), FSH (IU/L), testosterone (ng/L), Inhibine B (ng/L) and Insulin-like factor 3 (INSL3, ng/ml).
  Blood analyses will be repeated 3, 6, 9 and 12 months after the transplantation procedure.
Biomarker Study | Each patient in the study will be followed-up after screening during a period of 12 months post-grafting on 3, 6, 9 and 12 months after initial grafting.
  As an exploratory part of this study, the investigators will study the possibility to predict the presence of testicular spermatogenesis in a non-invasive way (by semen and/or urine samples). If different biomarkers could be identified specificaly for the different stages of spermatogenesis, the development of the transplanted biopsies could be monitored this way. For this study, a urine and semen sample will be needed 3, 6, 9 and 12 months after the transplantation procedure.
Complications | Each patient in the study will be follow-up after screening during a period of 15 months post-grafting.
  Each patient in the study will be followed-up during a period of 15 months after initial grafting or 3 months after graft-removal to report any complication(s) of the procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Vloeberghs, MD, Principal Investigator — CRG UZ Brussel
Locations (1):
- UZ Brussel Centre for Reproductive Medicine, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No